CLINICAL TRIAL: NCT06023420
Title: Using A Special 4 Herbs Formula For The Palliative Care Of Patients Suffering From Bone Secondaries
Brief Title: Efficacy of a Herbal Formula for Bone Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheng King Fai, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021.746-T
Record Dates: First submitted 2022-06-13; First posted 2023-09-05 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Herbal formula 5g daily, and Zometa
  Interventions: Drug: 4 Herbs Formula
- Control group (Active Comparator): Zometa alone
  Interventions: Drug: 4 Herbs Formula

INTERVENTIONS:
Drug: 4 Herbs Formula — 4 herbs formula dose: 5g/day
  Other Names: Zometa

SUMMARY:
RATIONALE: Nearly 50% of patients with bone metastases develop one or more complications collectively termed skeletal-related events (SREs). The study herbal medicine might reduce the morbidities due to "Skeletal-related events" (SRES), and extend survival time.

PURPOSE: the study is to explore the effects of the 4 Herbs Formula on the reduction of "Skeletal-related events" (SRES), and survival time.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Primary efficacy end points are SRE, general state and biomarkers. Secondary Survival rate and survival time Time to first SRE (since randomization) Biochemical markers Quality of Life: EQ5-D Pain control (Brief Pain Inventory)

OUTLINE:

Patients will be randomized to receive either 4 herbs formula plus Zometa or Zometa alone after all the eligibility criteria have been fulfilled and informed consent has been signed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Breast cancer bone metastasis-no supplementary treatment or hormonal treatment alone
* Confirmed diagnosis of metastatic breast cancer
* Radiographic proof of metastatic bone disease
* Informed consent obtained

Exclusion Criteria:

* Known history of primary bone tumors (benign and/or malignant)
* Prior use of bone modifying agents, including but not limited to zoledronic acid or denosumab within 12 months of study entry
* Active anti-cancer therapies in the form of cytotoxics or targeted therapies. [Patients who are currently on hormonal therapies, including but not limited to tamoxifen, aromatase inhibitors and LHRH agonists/antagonists are allowed for study entry. Clarifications shall be sought from investigators if in doubt].
* Significant drug hypersensitivity
* No informed consent signed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
reducing the morbidities of "Skeletal-related events" (SRES) extending survival time | 3 months
  SREs are defined as pathologic fractures, spinal cord compression, surgery to bone, radiation therapy to bone, and hypercalcemia of malignancy (HCM).

SECONDARY OUTCOMES:
Survival rate and survival time | Proportion of participants in all groups with overall survival at 1 year
  Proportion of participants in each group with overall survival at 6 months